CLINICAL TRIAL: NCT05792943
Title: Impact of Routine UGT1A1 Genotyping Before Irinotecan Chemotherapy in Taiwanese Cancer Patients
Brief Title: UGT1A1 Genotyping in Taiwanese Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202209008RINB
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-09

CONDITIONS: The Influence of the UGT1A1 Genotype

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Irinotecan is commonly used to treat lung, colorectal, pancreatic, stomach, esophageal, and other types of cancer. The main metabolic pathway of SN-38, the active product of Irinotecan, is grape glycoalkaloid acidification by UDP - glucuronosyltransferase (UGT1A1) and then excreted through bile and urine. Clinically, Irinotecan treatment can cause many adverse reactions, and differences in UGT1A1 genotypes can lead to structural changes or functional defects in enzymes, causing reduced acidification of grape glycolaldehyde, and increasing Irinotecan side effects. Therefore, if the patient's ability to metabolize the drug can be assessed before taking the drug, it will be of great help in treatment.

Until 2021, cancer will remain the top ten causes of death in Taiwan, of which colorectal and pancreatic cancer rank third and seventh among the top ten cancers in Taiwan, respectively, and these two cancers often use complex chemotherapy including irinotecan. Routine detection of UGT1A1 genotype in patients with colorectal and pancreatic cancer before irinotecan treatment predicts the drug metabolism capacity of irinotecan and adjusts the dose, allowing patients receiving irinotecan to reduce the harm of side effects. At present, the UGT1A1 genotype evaluated is usually only UGT1A1*28, but the common UGT1A1 genotype in Taiwan also has UGT1A1*6 and UG1A1*63, etc. There is no literature on Taiwanese cancer patients with actual irinotecan chemotherapy, so this study aims to explore the influence of the UGT1A1 genotype and develop other UGT1A1 genotype test methods. It is expected that molecular testing tools can improve cancer precision medicine and provide personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

Colorectal or pancreatic cancer patients.

Exclusion Criteria:

Age less than 20 or greater than 90.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of this project is patients with colorectal or pancreatic cancer from the National Taiwan University Cancer Center. A total of 100 cases are expected to be enrolled, ranging in age from 20 to 90 years old.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Using Sanger sequencing and real-time polymerase chain reaction analysis to study the distribution of UGT1A1 gene in cancer patients in Taiwan. | One month after receiving the samples.
  After Sanger sequencing and qPCR analysis, we classify several common types, such as UGT1A1*28, UGT1A1*6, and UGT1A1*63. Additionally, we aim to identify whether there are any other mutation points.

IPD SHARING:
Plan to Share IPD: No